CLINICAL TRIAL: NCT05140096
Title: An Open-Label, Fixed Sequence Study in Healthy Subjects to Assess the Pharmacokinetics of Acalabrutinib and Its Active Metabolite, ACP-5862, When Administered Alone and in Combination With Moderate CYP3A4 Inhibitors Fluconazole or Isavuconazole
Brief Title: A Study to Evaluate the Effect of Pharmacokinetics (PK) of Acalabrutinib and Its Active Metabolite (ACP-5862) When Administered Alone and With Moderate CYP3A4 Inhibitors Fluconazole or Isavuconazole in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-114
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy participants; Acalabrutinib; ACP-196, Active metabolite; ACP-5862; Fluconazole; Isavuconazole; CYP3A4 Inhibitors; Pharmacokinetics; PK; Safety
MeSH Terms: interventions — acalabrutinib; Fluconazole; isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment AB (Experimental): Participants will receive a single oral dose 100 mg acalabrutinib capsule on Day 1 of Period 1 (Treatment A) and later will receive single oral loading dose of 400 mg fluconazole tablets on Day 1, one hour prior to a single oral dose of 100 mg acalabrutinib in Period 2 (Treatment B).
  Interventions: Drug: Acalabrutinib; Drug: Fluconazole
- Treatment AC (Experimental): Participants will receive a single oral dose 100 mg acalabrutinib capsule on Day 1 of Period 1 (Treatment A), and later will receive oral dose of 200 mg iscavuconazole capsules three times daily (approximately every 8 hours apart) on Day 1, followed by 200 mg iscavuconazole capsule once daily from Day 2 to Day 5 with a single oral dose of 100 mg acalabrutinib capsule coadministered on Day 5 in Period 2 (Treatment C).
  Interventions: Drug: Acalabrutinib; Drug: Isavuconazole

INTERVENTIONS:
Drug: Acalabrutinib — Modify as "Participants will receive a single oral dose of 100 mg (1 X 100 mg capsule) acalabrutinib either on Day 1 of Period 1 (Treatment A) and Day 1 of Period 2 (Treatment B) or Day 5 of Period 2 (Treatment C).
Drug: Fluconazole — Participants will receive 400 mg fluconazole (2 × 200 mg tablets) on Day 1 Period 2 (Treatment B).
  Arms: Treatment AB
Drug: Isavuconazole — Participant will receive oral dose of 200 mg isavuconazole (2 × 186 mg of isavuconazonium sulfate capsules) three times daily on Day 1 and 200 mg isavuconazole (2 × 186 mg of isavuconazonium sulfate capsules) once daily on Days 2 to 5 in Period 2 (Treatment C).
  Arms: Treatment AC

SUMMARY:
This study will evaluate the effect of fluconazole and isavuconazole on the PK of acalabrutinib and its active metabolite, ACP-5862.

DETAILED DESCRIPTION:
This is a 2-period study. On Day 1 of Period 1, all participants will be randomized to 1 of 2 treatment sequences and will receive a single oral dose of 100 mg acalabrutinib (Treatment A). In Period 2, the participants who participated in Period 1 will receive either Treatment B (fluconazole) or Treatment C (isavuconazole). In Period 2 Treatment B, participants will receive a single oral loading dose of 400 mg fluconazole on Day 1 one hour before a single oral dose of 100 mg acalabrutinib. In Period 2 Treatment C, participants will receive oral dose of 200 mg isavuconazole three times daily (TID; approximately 8 hours apart) on Day 1 and 200 mg isavuconazole once daily (QD) from Day 2 to Day 5 with a single oral dose of 100 mg acalabrutinib coadministered on Day 5. There will be a washout of at least 8 days between Period 1 and first dose in Period 2. All participants will return to the study site approximately 7 days after the last study drug for follow-up procedures and adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker participant who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study
* Have body mass index of >= 18 kg/m^2 and <= 32 kg/m^2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the principal investigator (PI)
* Women participants must be of non-childbearing status and must have undergone the protocol specified sterilization procedures, and have official documentation, at least 6 months prior to the first dose; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone serum levels consistent with postmenopausal status
* Male participants must be willing to use protocol specified contraception methods
* Male participants must agree not to donate sperm from the first dosing until 90 days after the last dosing
* Ability to swallow multiple capsules and/or tablets using size 0 blank capsules (up to a maximum of 3 capsules per participant)

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* Presence of any clinically significant, ongoing systemic bacterial, fungal, or viral infections (including upper respiratory tract infections, but excluding localized cutaneous fungal infections), in the opinion of the PI
* History of any major surgical procedure within 30 days before the first dose of study drug
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing
* History or presence of clinically significant hypersensitivity or idiosyncratic reaction to acalabrutinib, fluconazole, isavuconazole, related compounds, or any inactive ingredients
* History or presence of liver disease and diabetes mellitus
* History of stroke or intracranial hemorrhage within 6 months before the first dosing
* History of bleeding diathesis
* Any clinically significant condition that may affect acalabrutinib absorption in the opinion of the PI, including gastric restrictions and bariatric surgery (eg, gastric bypass). Participants with cholecystectomy will be allowed.
* QTcF interval is >460 msec (males) or >470 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening
* Women who are pregnant or lactating
* Positive urine drug or alcohol results at screening or first check-in
* Positive urine cotinine at screening
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti-HBs), hepatitis B core antibody (anti-HBc), or hepatitis C virus (HCV)
* Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening
* Estimated creatinine clearance <90 mL/min and hemoglobin level below the lower limit of normal at screening
* Have been on a diet incompatible with the on-study diet, in the opinion of the PI, within the 28 days prior to the first dose of study drug, and throughout the study
* Donation of blood or significant blood loss within 56 days and plasma donation within 7 days prior to the first dose of study drug
* Unable to refrain from or anticipates the use of:

  * Any drugs, including prescription and nonprescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study
  * Any drugs known to be significant inducers or inhibitor of Cytochrome P450 (CYP) enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study, including drugs with a narrow therapeutic window that are P-gp substrates such as digoxin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve to the Last Observed Nonzero Concentration (AUC0-t) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Area Under the Plasma Concentration-time Curve to Infinity (AUC0-inf) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Maximum Observed Plasma Concentration (Cmax) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)

SECONDARY OUTCOMES:
Percent of Area Under the Plasma Concentration-time Curve to Infinity Extrapolated (AUC%extrap) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Time of the Maximum Observed Plasma Concentration (Tmax) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Time of the Last Measurable Nonzero Plasma Concentration (Tlast) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Apparent Terminal Elimination Half-life (T1/2) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Apparent Terminal Elimination Rate Constant (Kel) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Acalabrutinib | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Apparent Volume of Distribution During the Terminal Elimination Phase After Oral (Extravascular) Administration (Vz/F) of Acalabrutinib | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Metabolite-to-parent Molar Ratio for AUC0-t (MR_AUC0-t) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Metabolite-to-parent Molar Ratio for AUC0-inf (MR_AUC0-inf) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Metabolite-to-parent Molar Ratio for Cmax (MR_Cmax) of Acalabrutinib and ACP-5862 | Pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours post-acalabrutinib dose in each period (i.e., Days 1 to 2 for Treatments A and B and Days 5 to 6 for Treatment C)
Incidence of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through 30 days after the last dose of study drug (approximately 3. 5 months)
Incidences of Abnormal Vital Signs and Physical Examinations Reported as TEAEs | Day 1 through 30 days after the last dose of study drug (approximately 3. 5 months)
Incidences of Abnormal Electrocardiograms (ECGs) Reported as TEAEs | Day 1 through 30 days after the last dose of study drug (approximately 3. 5 months)
Incidences of Abnormal Clinical Laboratory Parameters Reported as TEAEs | Day 1 through 30 days after the last dose of study drug (approximately 3. 5 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home